CLINICAL TRIAL: NCT01329484
Title: Computerized Personal Interventions for Alzheimer's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Tzvi Dwolatzky, Mental Health Center, Beer-Sheva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-AD-TD-CTIL
Record Dates: First submitted 2011-03-30; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; Dementia; Computer; Cognitive training; Reminiscence therapy
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive training (Experimental)
  Interventions: Behavioral: Cognitive training
- Reminiscence therapy (Experimental)
  Interventions: Behavioral: Reminiscence therapy
- Control (Other): This group will receive neither of the above interventions or any other similar interventions
  Interventions: Other: No treatment

INTERVENTIONS:
Behavioral: Reminiscence therapy — Personalized reminiscence therapy using a computerized system
  Arms: Reminiscence therapy
Behavioral: Cognitive training — Cognitive training using a computerized system
  Arms: Cognitive training
Other: No treatment — Participants in the control group will receive neither of the 2 experimental interventions or any other similar interventions.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether the use of computerized systems in 2 common non pharmacological therapies (cognitive training and reminiscence therapy) will improve the cognitive function of patients with mild to moderate Alzheimer's disease (AD), or at least delay its deterioration. In addition, the investigators hypothesize that using the computerized systems will result in improved well-being of the patients and their main caregivers / family members, and in improved patient-caregiver and patient-family relations.

DETAILED DESCRIPTION:
Reminiscence therapy and cognitive training are two of the most common non-pharmacological therapies used to treat AD. To date, there is no clear evidence regarding the impact of these treatments on the cognitive function of people with AD. The inconclusive evidence may be due to methodological limitations, the availability of a limited number of controlled studies, the lack of standardized interventions and the need for sensitive assessment tools.

Increasingly, computerized systems are being designed to support both the cognitive assessment of patients with Alzheimer's disease and the administration of novel non-pharmacological interventions. Studies suggest that such systems may be of clear benefit. For example, in an initial study involving patients with AD, computerized cognitive training systems have been shown to be of value in providing a more standardized approach to cognitive training. Also, another study found that the use of a computerized system for reminiscence therapy was successful in facilitating patient-caregiver interaction.

Our research is a collaborative effort designed to test the effects of two such computer-supported interventions in patients with mild AD. The purpose of the research is to compare the efficacy of personalized computerized reminiscence therapy and that of computerized cognitive training to a control group. The reminiscence therapy program is based on developing an internet-based personalized reminiscence system, which will facilitate flexible interactive use by patients and caregivers. The importance of a personalized system is especially salient in immigrant, or in highly mobile, societies due to the heterogeneous background of the patients.

Separate preliminary studies have found positive effects of each system. The research will use various measures to evaluate the efficacy of both treatments, including the Mindstreams (NeuroTrax Corp., NJ) computerized neuropsychological assessment instrument, which will serve as the cognitive outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* MMSE score of 14-26

Exclusion Criteria:

* Visual impairment
* Auditory impairment
* Psychiatric disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive function measured by Mindstreams (NeuroTrax Corp., NJ) computerized neuropsychological assessment instrument. | baseline
Cognitive function measured by Mindstreams (NeuroTrax Corp., NJ) computerized neuropsychological assessment instrument. | Baseline+1 month
Cognitive function measured by Mindstreams (NeuroTrax Corp., NJ) computerized neuropsychological assessment instrument. | Baseline+3 months
Cognitive function measured by Mindstreams (NeuroTrax Corp., NJ) computerized neuropsychological assessment instrument. | Baseline+6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD, Principal Investigator — Mental Health Center, Beer-Sheva
Locations (2):
- Israel (2):
  - Mental Health Center, Beersheba
  - Memory Clinic, Shaare Zedek Medical Center, Jerusalem